CLINICAL TRIAL: NCT05593185
Title: Expanded Access Program (EAP) for Galinpepimut-S (GPS) in Patients Diagnosed With Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Brief Title: Expanded Access Program (EAP) for Galinpepimut-S (GPS) in Patients Diagnosed With AML or MDS
Status: Available | Type: Expanded Access
Sponsor: Sellas Life Sciences Group (Industry)
Responsible Party: Sponsor
Other Study IDs: SLSG22-401 EAP
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: blood cancer; blood-forming cells; bone marrow; Wilms Tumor-1 protein; immunizing therapy; hematological malignancies
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Hematologic Neoplasms

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Galinpepimut-S

SUMMARY:
Single patient expanded access program to provide galinpepimut-S for eligible patients with AML or MDS who have no other treatment option.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with AML or MDS, as assessed by their Treating Physician;
* Have no appropriate, comparable, or satisfactory alternative treatment available, or such alternatives have been tried without clinical success, including clinical studies;
* Inability to participate in a GPS clinical study for the disease or conditions; and
* Have a treating physician who has appropriately evaluated the benefit/risk profile for potential GPS treatment.
* Patients must have a diagnosis of either AML or MDS.
* Male or female patients > 18 years of age on the day of signing informed consent.
* Patients, or their legal representatives, must be able to communicate well with the Treating Physician, to understand and comply with the requirements for the provision of Expanded Access to GPS.
* Patients, or their legally acceptable representatives, must be willing and able to understand and provide signed informed consent for the EAP prior to the start of treatment that fulfills Institution Review Board (IRB) guidelines.
* Patients with AML must have had undergone SCT following morphological complete remission with or without peripheral blood (PB) counts recovery (CR/CRi). Patients with MDS are not required to have had CR prior to transplant.
* Patients with AML must have had Minimal Residual Disease (MRD) positivity per flow cytometry, RT PCR or NGS prior to SCT conditioning. Patients with MDS may have had less than CR prior to SCT. There is no requirement for specific SCT conditioning and conditioning intensity could have been myeloablative or nonmyeloablative (reduced intensity) conditioning.
* Patients must be consented within 30 -120 days after the date of SCT.
* Patients may concurrently be administered HMA +/- venetoclax and/or FLT3 ITD targeted agents at the discretion of the Treating Physician, in which case their regimen of GPS administrations will continue in parallel with the prescribed HMA +/- venetoclax and/or FLT3 ITD targeted agents regimen.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, 2 or 3.
* Patients must have an estimated life expectancy >6 months.
* If female, patients must be postmenopausal (at least 12 sequential months of amenorrhea) or surgically sterile. Females of childbearing potential must have a negative pregnancy test.
* Female patients of childbearing potential who are heterosexually active and male patients with female sexual partners of childbearing potential must agree to use an effective method of contraception (e.g., oral contraceptives, double-barrier methods such as a condom and a diaphragm, intrauterine device) during the GPS treatment and for 4 months following the last dose of GPS, or to abstain from sexual intercourse for this time; a woman not of childbearing potential is one who has undergone bilateral oophorectomies or who is post-menopausal, defined as the absence of menstrual periods for 12 consecutive months.
* Patients must not have end stage renal disease.
* Patients must have adequate hepatic function defined as a serum total bilirubin <2 × ULN (except for Gilbert'ssyndrome, which will allow bilirubin ≤3.0 mg/dL), and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 × ULN.
* Patients must be willing and able to return to the clinical site for adequate follow-up and to comply with the EAP treatment schedule, as required.

Exclusion Criteria:

* Prior clinically significant allergic reaction to Montanide, sargramostim (GM-CSF) or filgrastim (granulocyte colony stimulating factor [G-CSF]).
* Patients with acute promyelocytic leukemia (APL) or any morphologic and molecular variants, inclusive.
* Patients with a serious concurrent illness that in the opinion of the Treating Physician would pose an undue risk to the patient.
* Patients who currently have central nervous system leukemia.
* Patients who have received a live vaccine within 30 days prior to the first dose of EAP drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed. Vaccines used for the prevention of COVID-19 are allowed to be used as they are not live vaccines.
* Patients currently receiving systemic immunosuppressive therapy in dosing exceeding 10 mg daily of prednisone equivalent. The use of physiologic doses of corticosteroids or other immunosuppressive agents may be approved after consultation with the Sponsor. Steroids taken as short-term therapy (≤ 7 days) for antiemesis are permissible as are steroids with low systemic bioavailability (e.g., budesonide).
* Patients who have a known additional malignancy that is progressing or has required active treatment within the past 5 years, even if currently inactive or unapparent.
* Patients who have a known active CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during EAP screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of treatment.
* Patients who had a previous clinically significant systemic allergic reaction to Montanide, sargramostim (GMCSF), or filgrastim (G-CSF).
* Patients who have an active life-threatening infection requiring systemic therapy.
* Patients who have a history or current evidence of any condition, therapy, or laboratory abnormality that is not in the best interest of the patient to participate, in the opinion of the Treating Physician. This includes any serious, intercurrent, chronic, or acute illness, such as cardiac disease (New York Heart Association [NYHA] class III or IV), hepatic disease, or other illness considered by the Treating Physician as an unwarranted high risk for investigational drug treatment.
* Patients who have a known psychiatric or substance abuse disorder that would interfere with the patient's ability to cooperate with the requirements of the EAP.
* Patients who are pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the EAP, starting with the screening visit through 30 days after the last dose of EAP treatment.
* Patients who have had an allogeneic solid organ transplant.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult